CLINICAL TRIAL: NCT05846048
Title: Marital Rape:Knowledge, Attitudes and Prevalence in Asample of Married Women in Sohag Governorate
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Alaa Mohamed Mahmoud, principle investigator, Sohag University
Other Study IDs: Soh-Med-23-11-03MS
Record Dates: First submitted 2023-04-26; First posted 2023-05-06 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Marital Rape Knowledge ,Attitudes and Prevalence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: semi-structures questionaire — semi -structured questionnaire prepared by the researcher collect sociodemographic data , awareness ,attitudes about marital rape and health consequences

SUMMARY:
this study aims at estimation of prevalence of marital rape attitudes and knowledge towards it using semi structured questionnaire

DETAILED DESCRIPTION:
this study trying to estimate knowledge of married women in sohag about marital rape attitudes towards it the size of the problem psychological , mental ,physical health consequences if the problem deserve criminalization

ELIGIBILITY:
Inclusion Criteria:

* married or previously married females

Exclusion Criteria:

* mentally disabled or who with low IQ

Ages: 15 Years to 70 Years | Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: married females in sohag governorate
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
attitudes to marital rape questionnaire | 6 months
  married waomen know about marital rape or not

SECONDARY OUTCOMES:
prevalence of marital rape questionnaire | 6 months
  size of the proplem

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Basile KC. Prevalence of wife rape and other intimate partner sexual coercion in a nationally representative sample of women. Violence Vict. 2002 Oct;17(5):511-24. doi: 10.1891/vivi.17.5.511.33717. PMID 12477095
- [Background] Bergen RK, Bukovec P. Men and intimate partner rape: characteristics of men who sexually abuse their partner. J Interpers Violence. 2006 Oct;21(10):1375-84. doi: 10.1177/0886260506291652. PMID 16940402
- [Background] Jackson AL. State contexts and the criminalization of marital rape across the United States. Soc Sci Res. 2015 May;51:290-306. doi: 10.1016/j.ssresearch.2014.10.001. Epub 2014 Oct 14. PMID 25769868